CLINICAL TRIAL: NCT03485859
Title: Effect of Abdominal Binder aftEr Laparoscopic Treatment on Postoperative Recovery (BELT): a Randomized Controlled Trial
Brief Title: Effect of Abdominal Binder aftEr Laparoscopic Treatment on Postoperative Recovery
Acronym: BELT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Taejong Song, Professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-03-039
Record Dates: First submitted 2018-03-20; First posted 2018-04-02 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Laparoscopy
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): In subjects allocated to the abdominal binder group, the abdomen binder with a standard height of 22 cm (Sejung Korea, Seoul, Republic of Korea) was applied before leaving the operating room. The binder was placed on the abdomen across the laparoscopic incision, with the upper border not higher than the lower margin of the rib cage, ensuring minimal restriction of lateral costal expansion and diaphragmatic excursion. Subjects were carefully instructed to use the abdominal binder during at least the first 2 consecutive days and night, and to reposition the abdominal binder correctly when needed.
  Interventions: Device: Experimental group
- Control group (Placebo Comparator): In subjects allocated in the control group, subjects were not given any opportunity to ware an abdominal binder.
  Interventions: Device: Control group

INTERVENTIONS:
Device: Experimental group — In subjects allocated to the abdominal binder group, the abdomen binder with a standard height of 22 cm (Sejung Korea, Seoul, Republic of Korea) was applied before leaving the operating room. The binder was placed on the abdomen across the laparoscopic incision, with the upper border not higher than the lower margin of the rib cage, ensuring minimal restriction of lateral costal expansion and diaphragmatic excursion. Subjects were carefully instructed to use the abdominal binder during at least the first 2 consecutive days and night, and to reposition the abdominal binder correctly when needed.
  Arms: Experimental group
Device: Control group — In subjects allocated in the control group, subjects were not given any opportunity to ware an abdominal binder.
  Arms: Control group

SUMMARY:
There have been no studies exploring the efficacy of incision support using an elastic abdominal binder after laparoscopy to date. The investigators performed therefore a randomized controlled trial to determine the effect of post-laparoscopic abdominal binder use on enhanced recovery after surgery (ERAS) in patients with gynecologic disease.

DETAILED DESCRIPTION:
An abdominal elastic binder (girdles, trusses, abdominal belts, longuette, etc.) is a wide belt that surrounds the abdomen and supports the incision . Abdominal binder is routinely used after open surgery and Cesarean section, because it has been reported, according to a recent systematic review, to facilitate enhanced recovery after surgery (ERAS) such as pain relief, reduced risk of seroma formation, improved respiratory function, and assisted physical function using additional support to the lower abdominal musculature.

However, the routine use of abdominal binder after laparoscopy has been challenged due to a potential risk of postoperative pulmonary complications and deep venous thrombosis due to increased intra-abdominal pressure. Also, abdominal binders after laparoscopy have been criticized for being uncomfortable and hot to wear and for impinging the breast line in females. Therefore, some laparoscopists prefer the use of abdominal binder in patients undergoing laparoscopy, while other laparoscopists did not. However, there have been no studies exploring the efficacy of incision support using an elastic abdominal binder after laparoscopy to date. The investigators performed therefore a randomized controlled trial to determine the effect of post-laparoscopic abdominal binder use on ERAS in patients with gynecologic disease.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years
* American Society of Anesthesiologists physical status (ASAPS) classification I-II
* absence of pregnancy at the time of surgery

Exclusion Criteria:

* body mass index (BMI) ≥30 kg/m2
* history of abdominal surgery within 6 months
* history of ventral or incisional hernia
* walking disabilities (or walking with the assistance of crutches or a walker)
* chronic obstructive respiratory disease
* stage IV cancer,
* chronic pain syndrome (defined as daily intake of opioids for chronic back pain, chronic headache, or fibromyalgia)
* inability to fill out the questionnaire

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2018-08-05 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
postoperative pain | at 48 hours after surgery
  Subjects rated postoperative pain intensity using a visual analog scale (VAS) at 12, 24, and 48 hours after surgery. The scale was presented as a 10-cm line with verbal descriptors ranging from "no pain" to "worst imaginable pain".

SECONDARY OUTCOMES:
limitation of walking ability | at 48 hours after surgery
  Subjects were instructed to place a mark on a 10-cm line corresponding to the percentage of full-walking ability, with 0 cm representing no activity limitation and 10 cm being the maximal activity limitation.
Incentive spirometry performance | at 24 hours after surgery
  Volumetric incentive spirometry (Hyupsung Medical Co., Ltd, Yangju, Republic of Korea) was performed in all subjects at 24 hours after surgery, because inspiratory spirometry can be used as a simple mean to follow lung volume, especially vital capacity and inspiratory reserve volume, in postoperative period in spontaneous breathing patients.

CONTACTS AND LOCATIONS:
Overall Officials: Taejong Song, MD PhD, Principal Investigator — Kangbuk Samsung Hospital, Seoul, Republic of Korea
Locations (1):
- Kangbuk Samsung Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: No